CLINICAL TRIAL: NCT03658993
Title: Rifaximin-treatment of Collagenous Colitis:
Brief Title: Rifaximin-treatment of Collagenous Colitis
Acronym: XiCoCo
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bonderup, Ole K., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BonderupO
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Collagenous Colitis
Keywords: Microscopic colitis; Diarrhoea; Microbiome; Rifaxamine
MeSH Terms: conditions — Colitis, Collagenous; Colitis, Microscopic; Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: A prospective, randomised, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation and labelling follow guidelines defined by the Danish Medicines Agency and will be performed by the Hospital Pharmacy Region Midtjylland Clinical Trial Unit, Aarhus University Hospital and Norgine. For equal allocation to the two treatment arms computer generated block randomisation (blocks of 8) will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaxamine 550 mg (Active Comparator): Study drug Oral Rifaximin 550 mg TID for 4 weeks .
  Interventions: Drug: Rifaximin 550 MG
- Placebo (Placebo Comparator): Placebo TID for 4 weeks
  Interventions: Drug: Rifaximin 550 MG

INTERVENTIONS:
Drug: Rifaximin 550 MG — Oral Rifaximin 550 mg TID for 4 weeks.
  Other Names: Xifaxan

SUMMARY:
The hypothesis of this study is that an altered gut microbiota is a contributory factor in initiating an inflammatory process in the colonic mucosa leading to collagenous colitis. The investigators suggest that treatment with budesonide reduces the inflammation without treating the underlying cause. In this trial the investigators will try to modullate gut microbiota by adding rifaximin. The aim of this study is to assess if 4 weeks treatment with rifaximin as a supplement to a standard course of budesonide against active CC can reduce the risk of relapse after treatment cessation.

DETAILED DESCRIPTION:
Patients with biopsy-verified CC and active disease defined by >3 bowel movements/day or >1 watery stool measured as a mean for a week. Patients will be invited to participate in the study independently of age and disease duration.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent

  * Histological findings fulfill criteria for CC:

    * A subepithelial collagenous band >10 μm in colonic biopsies
    * Increased count of inflammatory cells in lamina propria
  * Diagnostic biopsies are a maximum of two years old
  * A history of nonbloody, watery diarrhea for more than two weeks prior to screening in patients with recently diagnosed CC or a history of clinical relapse for more than a week in patients with known CC
  * Active disease: > 3 stools/day or >1 watery stool/day measured as a mean during a week prior to baseline

Exclusion Criteria:

* - Significant findings at colonoscopy that could cause diarrhea (colonic diverticulosis and polyps < 2 cm are not considered significant findings)
* Biopsies more than two years old in a patient, who does not accept a new sigmoidoscopy
* Untreated celiac disease
* Positive stool cultures for pathogenic intestinal bacteria including Clostridium difficile
* Suspected colitis induced by medication (diarrhea shortly after commencement of NSAID's, statins, SSRI or PPI)
* Severe comorbidity (cardiovascular, renal, endocrine, neurologic, pulmonal or psychiatric) or history of cancer during the last 5 years
* Abnormal liver biochemistry (ALAT or ALP > 2,5 x upper limit), cirrhosis or portal hypertension
* Pregnancy or lactation (assured by negative P-hCG at inclusion)
* History of significant intestinal resection
* Treatment with 5-ASA, Salazopyrin, immunemudulators (Azathioprine, 6-mercaptopurine or Methotrexate), biologic drugs (TNF-alfa-inhibitors), local or systemic glucocorticoids (except for Budesonide) within the last three month
* Allergy or intolerance to Rifaximin (or similar antibiotics such as Rifampicin or Rifabutin)
* Expectation of lack of cooperation or insufficient comprehension
* Concomitant participation in an other clinical trial or participation within the last 30 days
* Patients receiving Warfarin or Marcoumar (interaction with risk of uncontrolled INR-levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | The number of patients in clinical remission 12 weeks after randomisation
  The number of patients in clinical remission in the Rifaximin group compared to the placebo group.

SECONDARY OUTCOMES:
Time to relapse. | Last visit is one year after treatment cessation.
  Time to relapse after cessation of treatment with Rifaxamin compared to placebo
Difference in Quality of life: short health scale (SHS) | 12 weeks after treatment
  Difference in Quality of life assessed by a visual analog scale (SHS) after cessation of treatment with Rifaxamin compared to placebo. The scale extends from 0 to 10 with 0 as worst outcome and 10 as best outcome.
Microbioma | 12 weeks after treatment
  Changes is gut microbiome after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabine K Becker, MD, Principal Investigator — Clinic of Gastrointestinal- and Infectious Diseases, Diagnostic Center Silkeborg Regional Hospital, Falkevej 1-3, 8600 Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of study completion
Access Criteria: Requestors will be required to sign a Data Access Agreement